CLINICAL TRIAL: NCT01509001
Title: Study of Metabolic and Haemodynamic Effects of Metformin and Glimepiride in Patients With Type 2 Diabetes
Brief Title: Study of Metabolic and Haemodynamic Effects of Metformin and Glimepiride in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria Elizabeth Rossi da Silva, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SILVAMER; CUNHAMR (Other: University of Sao Paulo)
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; metformin; glimepiride; glucose control; vascular reactivity; Adverse Reaction to Other Drugs and Medicines
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin (Active Comparator): Participants will randomized into Metformin (750 to 2500 mg/day) or Glimepiride (1 to 8 mg/day) therapy. After 4 months, the patients will crossed-over with no washout period to the alternative treatment for an additional 4-month period on similar dosage schedule
  Interventions: Drug: Metformin
- glimepiride (Active Comparator): Participants will randomized into Metformin (750 to 2500 mg/day) or Glimepiride (1 to 8 mg/day) therapy. After 4 months, the patients will crossed-over with no washout period to the alternative treatment for an additional 4-month period on similar dosage schedule
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Metformin — 750 to 2500 mg/day, two times a day during 4 months
  Other Names: glifage
  Arms: metformin
Drug: Glimepiride — 1 to 8 mg/day , two times a dya, during 4 months.
  Other Names: Amaryl
  Arms: glimepiride

SUMMARY:
Aim:

The purpose of this study is to compare the effects of glimepiride(G) and metformin(M) on vascular reactivity, haemostatic factors and glucose and lipid profile in patients with type 2 diabetes.

Methods:

A prospective study will be performed in 20 uncontrolled patients previously treated with dietary intervention. Participants will randomized into M (750 to 2500 mg/day) or G (1 to 8 mg/day) therapy. After 4 months, the patients will be crossed-over with no washout period to the alternative treatment for an additional 4-month period on similar dosage schedule.

* The following variables were assessed before (basal values) and after 4 months of each treatment period:

  1. Hormonal and metabolic determinations: fasting plasma glucose, insulin, catecholamine, lipid profile and HbA1 levels.
  2. Haemostatic factors: t-PA antigen and activity, PAI-1 antigen and activity, platelet aggregation, fibrinogen and plasminogen levels.
  3. Cardiovascular evaluation: flow indexes of carotid and brachial arteries. Also, at the end of each treatment period, a 12-hour metabolic profile including measurements of glucose, insulin, glucagon, proinsulin and triglycerides levels at fasting and every 2 hours (7:00 am to 7:00 pm)will be done

DETAILED DESCRIPTION:
Measurements were be made at fasting

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes patients with fasting glucose values >7.78 mmol/L and/or glycated hemoglobin exceeding 1.0% or more the normal range (4-8.5%) after 2 or more months of a diet therapy

Exclusion Criteria:

* any severe concomitant illness
* nephropathy (serum creatinine >1.6 mg/dL and microalbuminuria)
* uncontrolled hypertension (BP >190x120 mmHg)
* stroke
* peripheral vascular disease
* marked dyslipidemia (total cholesterol>6.5mM/L and triglycerides levels >2.8mM/L)
* coagulopathy
* proliferative retinopathy and use of hypolipemic and anticoagulant medications or autonomic neuropathy
* assessed by blood pressure response to standing
* beat-to -beat heart rate variation
* Valsalva maneuver and handgrip test.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
glucose control | every 2 weeks
  measurements of glucose , glycated haemoglobin and insulin levels

SECONDARY OUTCOMES:
haemodynamic improvement | every 4 months
  flow indexes of carotid and brachial arteries

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elizabeth R Silva, Md,Phd, Principal Investigator — University of Sao Paulo
Locations (1):
- Clinical Hospital of São Paulo Medical School, São Paulo, São Paulo, Brazil